CLINICAL TRIAL: NCT01110031
Title: An Open-Label, Single-Arm, Phase I Study to Evaluate the Effect of Ofatumumab on Cardiac Repolarization (QTc Duration) in Patients With Fludarabine-Refractory B-cell Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab Cardiac Repolarization (QTc) Study in Fludarabine-Refractory Chronic Lymphocytic Leukemia Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112855
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: Chronic lymphocytic leukemia; Cardiac Repolarization (QTc)
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Six months treatmet with ofatumumab will be given to subjects with chronic lymphocytic leukemia.
  Interventions: Biological: Ofatumumab

INTERVENTIONS:
Biological: Ofatumumab — Anti-CD20 monoclonal antibody
  Other Names: Arzerra

SUMMARY:
Ofatumumab is a fully-human monoclonal antibody that exhibits high binding affinity to an antigen on the surface of B lymphocytes. Antigen engagement by ofatumumab results in maximal B-cell killing through complement-dependent cytotoxicity and antigen-dependent cellular cytotoxicity in both antigen high- and low-expressing cells. Recent research has shown that ofatumumab-dependent B-cell depletion provides clinical benefit to subjects with CD20-positive cancers such as chronic lymphocytic leukemia (CLL). The purpose of the current study is to assess the impact of ofatumumab on electrocardiographic parameters with particular focus on cardiac repolarization (QTc interval duration) in subjects with refractory CLL. Subjects enrolled in this open-label, single-arm trial will receive ofatumumab at the highest clinical dose (2000 mg) studied or planned for study. Ofatumumab will be administered as eight weekly intravenous (IV) infusions followed by four monthly infusions, beginning in Week 13, across a 25-week treatment period. Cardiovascular effects will be evaluated during treatment through routine 12-lead electrocardiographic (ECG) monitoring. The pharmacokinetic relationship between plasma concentration of ofatumumab and its effect on QTc interval duration will be examined. Specifically, ECG assessments will be collected in triplicate at baseline, at the time of maximum ofatumumab concentrations periodically on-therapy, and at the end of treatment. After completion of the final ofatumumab infusion, subjects will continue to be followed for safety and efficacy for six months relative to the last ofatumumab dose.

DETAILED DESCRIPTION:
The purpose of this trial is to assess the impact of ofatumumab on electrocardiographic parameters with particular focus on cardiac repolarization (QTc interval duration) in subjects with refractory Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL).
* Active CLL disease and indication for treatment.
* Previous treatment with fludarabine-containing treatment that did not achieve at least a partial response or, disease progression occurred in responders within six months of the last dose of a fludarabine-containing treatment regimen.
* Fully active at a minimum, or fully capable of self-care and up and about more than 50% of waking hours.
* Age 18 years or older.
* Signed written informed consent.
* Acceptable levels of laboratory chemistry tests of potassium and magnesium.
* Males and female subjects must agree to use contraception (if fertile) from the time of the first dose of study medication until one year following last dose of ofatumumab.

Exclusion Criteria:

* Any abnormal electrocardiogram (ECG) or cardiac conduction findings .
* Certain heart problems, chronic infections, or serious significant diseases.
* Known transformation of CLL.
* CLL central nervous sytem involvement.
* Abnormal/inadequate blood values, liver, or kidney function.
* Past or current malignancy besides CLL, unless you have been free of malignancy for at least two years, have a history of completely resected non-melanoma skin cancer, or have been successfully treated.
* Lactating women or women with a positive pregnancy test.
* Use of medications known to prolong the heart rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05-13 (Actual); Primary Completion 2012-04-12 (Actual); Study Completion 2012-06-26 (Actual)

PRIMARY OUTCOMES:
Cardiac Repolarization (Fredericia's QTc) | 25-week ofatumumab treatment period
  ECGs are collected in triplicate during the study to assess QTc effect.

SECONDARY OUTCOMES:
Plasma concentrations of ofatumumab and electrocardiogram (ECG) parameters | 25-week ofatumumab treatment period
  The pharmacokinetic results will be correlated to ECG findings to determine if drug concentrations relate to any ECG effects.
Vital signs, weight, adverse events | 25-week ofatumumab treatment period plus 6-month follow-up after final ofatumumab infusion
  Safety and tolerability of ofatumumab therapy will be determined by analysing changes in vital signs, weight, or development of adverse events.
Flow cytometry | 25-week ofatumumab treatment period plus 6-month follow-up after final ofatumumab infusion
  Efficacy of ofatumumab therapy will be measured by the number of CD20 positive cells in the blood
Cytokine, chemokine, human anti-human antibodies | 25-week ofatumumab treatment period plus 6-month follow-up after final ofatumumab infusion
  Effect of ofatumumab on circulating biomarkers in refractory Chronic Lymphocytic Leukemia (CLL) subjects will be determined by measuring changes in the cytokine, chemokine, human anti-human antibody levels.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, La Jolla, California, United States
- GSK Investigational Site, Randwick, New South Wales, Australia
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch

REFERENCES:
- [Derived] Jewell RC, Laubscher K, Lewis E, Fang L, Gafoor Z, Carey J, McKeown A, West S, Wright O, Sedoti D, Dixon I, Hottenstein CS, Chan G. Assessment of the effect of ofatumumab on cardiac repolarization. J Clin Pharmacol. 2015 Jan;55(1):114-21. doi: 10.1002/jcph.376. Epub 2014 Aug 21. PMID 25103870
- See also: Results for study 112855 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112855?search=study&study_ids=112855#rs